CLINICAL TRIAL: NCT03979690
Title: A Pilot, Prospective, Non-randomized Study to Evaluate the Safety and Feasibility of Novel Single Use Robotic Colonoscopy System ("NISInspire-C System") in Human Subjects
Brief Title: Feasibility Study of a Novel Single Use Robotic Colonoscopy System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bio-Medical Engineering (HK) Limited (Industry)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NISInspire-001; HKUCTR-2616 (Registry Identifier: HKU Clinical Trials Registry (HKUCTR)); HKUCTR-2617 (Other: HKU Clinical Trials Registry (HKUCTR))
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Colonic Polyp; Colon Adenoma; Colorectal Cancer
Keywords: Robotic Colonoscopy; Tandem Colonoscopy; NISInspire-C System; Single Use Colonoscope; Colonoscopy
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects Receiving Colonoscopy (Experimental): Subjects receiving tandem colonoscopies using the NISInspire-C System followed by a Conventional Colonoscopy
  Interventions: Device: NISInspire-C System

INTERVENTIONS:
Device: NISInspire-C System — The NISInspire-C System is a disposable robotic colonoscopy system that consists of a flexible slender insertion tube designed to ensure non-invasive, reliable and safe colorectal screening. It comprises of two components: NISInspire-C Console, and the NISInspire-C Disposable Colonoscope.

SUMMARY:
This is a single centre, non-randomized, tandem colonoscopy trial of the NISInspire-C System, followed immediately by a conventional colonoscope (CC). Each trial subject will undergo colonoscopy using the NISInspire-C system, followed immediately by CC. The purpose of this study is to obtain observational data on the safety profile, feasibility and usability of the NISInspire-C System in performing diagnostic colonoscopy in human subjects. The level of procedural pain experienced by subjects will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 40 and 70 years, inclusive, at the time of informed consent
* Females aged between 55 and 70 years, inclusive, at the time of informed consent (Rationale: to include only women with non-childbearing potential to avoid completely pregnant trial subjects)
* Symptomatic adults indicated for elective colonoscopy, or asymptomatic adults willing to undergo a colonoscopic screening for polyps or colorectal cancer
* Adults without prior colonoscopy
* Able to provide a written informed consent form approved by an Independent Ethics Committee (IEC)/ Institutional Review Board (IRB), prior to any study-specific procedures
* Willing and able to comply with the study procedures

Exclusion Criteria:

* History of colorectal cancer, inflammatory bowel disease, polyposis syndrome, familial polyposis coli, hereditary nonpolyposis colorectal cancer syndrome, active diverticulitis or toxic megacolon
* Lower gastrointestinal bleeding within 28 days prior to the colonoscopy day
* Known bleeding tendency
* Received antiplatelet or anticoagulation therapy within 3 days prior to the colonoscopy day
* Known colonic stricture
* Known multiple sigmoid colon diverticula
* History of any abdominal or pelvis surgical procedures including colonic and rectal surgical resection
* Known abdominal wall hernias
* History of radiotherapy to the abdomen or pelvis
* Known coronary ischemia or cardiovascular stroke within 3 months prior to the colonoscopy day
* Contraindication to the proposed anaesthesia
* Received any investigational medicine or treatment within 28 days prior to Screening
* Any condition, in the opinion of the Investigator, that is unstable and could jeopardize the safety of the subject and their compliance in the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males Aged between 40 and 70 years; Females Aged between 55 and 70 years
Enrollment: 20 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of Intra-Operative and Post-Operative Adverse Events | 10 Days
  Number of Adverse Events
Feasibility: Caecal Intubation Rate (CIR) | 1 Hour
  CIR: Number of Times Caecum is Reached
Feasibility: Time-to-Caecum (TTC) | 1 Hour
  TTC: Time to Reach Caecum
Feasibility: Polyp Detection Rate (PDR) | 1 Hour
  PDR: Number of Polyps Detected

SECONDARY OUTCOMES:
Usability | Day 1 (Day of Procedure)
  Feedback on General Usage of the NISInspire-C Disposable Colonoscope

OTHER OUTCOMES:
Intra-Procedural Pain (Exploratory Outcome) | Day 1 (Day of Procedure)
  The Level of Procedural Pain Experienced by Subjects Undergoing the Colonoscopy Procedures will be Explored.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Keung Leung, Professor, Principal Investigator — Division of Gastroenterology & Hepatology, Department of Medicine, The University of Hong Kong, Queen Mary Hospital; Dominic Chi Chung Foo, Dr, Principal Investigator — Division of Colorectal Surgery, Department of Surgery, The University of Hong Kong, Queen Mary Hospital
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong